CLINICAL TRIAL: NCT06620315
Title: Comparison Between Primary and Secondary Implant Stability of Hybrid Versus Resorbable Blast Media (RBM) Surfaces Using Resonance Frequency Analysis
Acronym: IMPLANTSTABIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, RANA AHMAD, ASSISTANT PROFESSOR, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CPSP/REU/DSG-2018-262-2439
Record Dates: First submitted 2024-08-15; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Implant Complication; IMPANT STABILITY

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hybrid (sand blasted acid etched implants) (Active Comparator)
  Interventions: Combination Product: sand blasted implant
- RBM (Active Comparator): RBM implant
  Interventions: Combination Product: RBM

INTERVENTIONS:
Combination Product: RBM — Resorbable Blast Media (RBM) implant surfaces can enhance osseointegration and implant stability
  Arms: RBM
Combination Product: sand blasted implant — sand blasted implant
  Arms: Hybrid (sand blasted acid etched implants)

SUMMARY:
• To compare primary stability (during initial loading of implant) and secondary stability (after 12 weeks of implant loading) which are denoted as ISQ value of Hybrid (DIO UFII) versus Resorbable blast media (RBM) (Osstem TSII) implant surfaces.

DETAILED DESCRIPTION:
An approval from the hospital ethical committee will be obtained for this study. As a protocol all patients presenting to Institute of Dentistry, CMH Lahore Medical College will be examined in general OPD and those patients who fulfill the inclusion and exclusion criteria will be referred to Prosthodontics department. After history, complete oral examination and informed consent. Patients will be divided into two groups by lottery method; In Group 1 Hybrid (sand blasted acid etched implants) will be place. In Group 2 Resorbable Blast Media (RBM) implant surfaces will be placed. On the basis of randomized study the patients will be selected for the study to measure implant primary stability with a resonance frequency analyzer at the time of initial loading of implant, starting with an assessment immediately following implant placement with insertion torque of 30 Ncm and then secondary stability at 12 weeks post operatively by using Ostell Mentor. This instrument on each implant by inserting a standardized abutment (Smartpeg) of fixed length into each implant. The transducer probe (Osstell mentor probe) will be held so that the probe tip was aimed at the small magnet on top of the Smartpeg at a distance of 2-3 mm in both the buccal and lingual directions, and the mean of these measurements will then be calculated. The probe will be held still during the pulsing time until the instrument beeped and the displayed the ISQ value. ISQ1 will be evaluated immediately during initial implant loading which will be primary stability and ISQ2 will be evaluated after 12 weeks of implant placement when implant is properly osseointegrated, which will be secondary stability of an implant.

The implant fixtures will be DIO UF II for the Hybrid implants and the Osstem TSII plus system for the RBM implants. Data would be stratified for age, gender and implant site to address the effect modifiers.

ELIGIBILITY:
Inclusion Criteria:

* o Age between 20 to 50 years.

  * Both male and female patients will be selected.
  * Patients suitable for implant restorations on CBCT will be diagnosed by;

    1. Bone height (minimum of 12mm)
    2. Bone width (minimum of 5mm)
    3. Proximity with vital structures (nerves, blood vessels)

Exclusion Criteria:

* o Patients with diabetes, Parkinson's disease, myasthenia gravis and bulbar palsy

  * Diseases with either a strong connection to emotional stress or impairing mental health like depression, anxiety, sleeping disorder on history examination.
  * Patients with poor oral hygiene.
  * Patients with parafunctional habits of severe clenching habit, bruxism.
  * Heavy smokers
  * Patients who had undergone radiotherapy or chemotherapy.
  * Patients with osteoarthritis, osteoporosis.
  * Patients taking bisphosphonates

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Primary Stability | up to 3 months
  absence of clinically detectable implant mobility

SECONDARY OUTCOMES:
Secondary Stability | 3 months
  absence of clinically detectable implant mobility

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prosthodontics, Institute of Dentistry/CMH Lahore Medical College., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided